CLINICAL TRIAL: NCT01611194
Title: Brain Injury and Mechanisms of Action of HBO2 for Persistent Post-Concussive Symptoms After Mild Traumatic Brain Injury (BIMA) Protocol
Brief Title: mTBI Mechanisms of Action of HBO2 for Persistent Post-Concussive Symptoms
Acronym: BIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: S-11-17
Record Dates: First submitted 2012-05-03; First posted 2012-06-04 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Traumatic Brain Injury With Brief Loss of Consciousness; Post-Concussion Syndrome
Keywords: HBO2; HBOT; mTBI; Brain injury; PCS; PTSD; hyperbaric oxygen
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Injuries; Stress Disorders, Post-Traumatic | interventions — Oxyhemoglobins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBO2 at 1.5 Atomspheres Absolute (ATA) (Experimental): Hyperbaric oxygen (HBO2) at 1.5 atms. Stratified by site and time from injury (less than one year versus one year or more), in which participants are randomized. Each participant will complete 40 sessions, one session per day, five sessions per week, within 12 weeks following randomization.
  Interventions: Drug: Hyperbaric oxygen (HBO2) at 1.5 atms
- Sham Control (1.2 Atomspheres) (Sham Comparator): Sham control 1.2 atms. Each participant will complete 40 sessions, one session per day, five sessions per week, within 12 weeks following randomization. Breathing air at a pressure of 1.2 atm abs is equivalent to inhaling 25% oxygen at sea level pressure (1.0 atm abs).
  Interventions: Drug: Sham control 1.2 atms

INTERVENTIONS:
Drug: Hyperbaric oxygen (HBO2) at 1.5 atms — The Hyperbaric oxygen (HBO2) at 1.5 atms (active) group (hyperbaric oxygen-chamber compressed to 1.5 atm abs and breathing 100% oxygen). Each participant should complete 40 sessions over the course of 12 weeks, one session per day, five per week.
  Other Names: 1.5 atms
  Arms: HBO2 at 1.5 Atomspheres Absolute (ATA)
Drug: Sham control 1.2 atms — The chamber will be compressed with air to 1.2 atm abs to simulate the active group. Participants will don a hood and breathe 21% oxygen (room air). Each participant will complete 40 sessions, one session per day, five sessions per week, within 12 weeks following randomization. Breathing air at a pressure of 1.2 atm abs is equivalent to inhaling 25% oxygen at sea level pressure (1.0 atm abs).
  Other Names: 1.2 atms (shame)
  Arms: Sham Control (1.2 Atomspheres)

SUMMARY:
Purpose of this study is to investigate the mechanisms of action of hyperbaric oxygen therapy for persistent post-concussive symptoms after mild tramatic brain injury

DETAILED DESCRIPTION:
Active duty military personnel and Veterans received for 60-minute daily chamber sessions in which they received HBO2, 1.5 atmospheres absolute (ATA), or sham intervention (1.2 ATA, room air) for post concussion syndrome (PCS).

The study is to provide a rationale for the selection of outcome assessments to serve as primary and secondary endpoints for a pivotal randomized clinical trial of hyperbaric oxygen for the treatment of PCS. The participants will undergo a comprehensive battery of symptom and quality of life assessments. The distribution of response, change in response over time, homogeneity of variance across subgroups, and relationships between outcome measures will be compared by treatment assignment with a cohort from a study of similar design among a normal study population.

ELIGIBILITY:
Inclusion Criteria

* On active duty (TRICARE beneficiary) at the time of consent and through the 6-month visit or a Veteran, as well as Active Duty military who become Veterans after enrollment.
* Men and women 18-65 years of age at the time of study enrollment.
* Able to equalize middle ear pressure in a test of chamber pressure and tolerate the chamber environment.
* Able to speak and read English, as primary language.
* Agrees to and appears able to participate in all outcome assessments.
* Agrees to provide blood samples for clinical lab tests.
* Demonstrates the ability to offer informed consent and signs the study informed consent document.
* Participants stationed or living outside the Colorado Springs/Denver, Colorado area must be willing and able to travel. A reliable companion may accompany the participant if travel supervision is required.
* Active duty participants must obtain a letter of support from a supervisor or commanding officer prior to the outcome assessments (and travel, if necessary) to the OAC.

Participants must have a history of at least one (minimum requirement) mild traumatic brain injury (mTBI) with persistent symptoms that meets all the following criteria:

* Brain injury that occurred more than 3 months prior to baseline screening at the local site, with the most recent injury occurring no more than 5 years prior to randomization.
* Most recent traumatic brain injury (TBI) occurred on active duty.
* TBI was caused by non-penetrating trauma or blast exposure.
* TBI resulted in at least one of the following at the time of injury: a period of loss of or a decreased level of consciousness (up to 30 minutes); a loss of memory for events immediately before or after the injury (up to 24 hours); or alteration in mental state at the time of the injury (becoming dazed or confused).
* Has current complaints of TBI symptoms such as headache, dizziness, or cognitive or affective problems that score at least 3 post-concussive symptoms as assessed by the OSU TBI-ID.
* Has received current standard of care pharmacologic and nonpharmacologic interventions for TBI and any concomitant post traumatic stress disorder (PTSD) with no significant change in psychoactive therapy for at least 1 month.
* Creatinine level that is less than or equal to the EACH laboratory's upper limit of normal. If the creatinine level exceeds the EACH laboratory's upper limit of normal, participants cannot have a CT scan due to risk of contrast dye-induced renal failure. Such participants may be randomized but must be approved by the Study Director.

Exclusion Criteria:

* Prisoners.
* Pregnant Women.
* Minors.
* Individuals whose most recent TBI was sustained during illegal activity.
* Potential active duty participants stationed >1 hour outside the designated recruitment area of a participating local site will be excluded unless the command authorizes temporary relocation and appropriate relocation resources.
* Potential Veteran participants who live >1 hour outside the designated recruitment area of a participating local site, must be willing and able to travel to the local site to participate in all required local site visits without additional financial assistance than that which is described in the Veteran Payment Schedule (consent attachment C).
* Active duty individuals with anticipated prolonged TAD/TDY or deployment within 6 months of study enrollment will be excluded.
* Veterans with anticipated prolonged travel or relocation within 6 months of study enrollment will be excluded.

An individual with any of the following characteristics will be excluded from this study based on contraindications to hyperbaric pressurization and hyperbaric oxygenation or other study assessment measures:

* Women who are pregnant or who plan to become pregnant during the study period.
* Women who are breastfeeding.
* Women of childbearing potential who do not agree to practice an acceptable form of birth control during the study period.
* Epilepsy or seizure disorder not stable on anticonvulsant therapy (stable defined as 6 months seizure-free).
* Inability to protect airway or requires frequent suctioning.
* Known or suspected perilymphatic fistula.
* Presence of tracheostomy (due to limitations in autoinflation of the middle ear space).
* Diabetes (risk of hypoglycemia).
* Creatinine level that exceeds 1.5 times the EACH laboratory's upper limit of normal.
* A diagnosis (from patient report or medical record evidence within one year) of untreated clinical hypo- or hyperthyroidism.
* Allergy to iodine-based contrast dye (exclusion criteria for neuroimaging assessment measures only).
* Presence of implanted device (e.g., cardiac defibrillator, intrathecal drug delivery device, cochlear implant, pacemaker, stents or aneurysm clips) that poses increased risk to the participant during hyperbaric exposure or magnetic resonance imaging (MRI). Any implanted device must be cleared through the manufacturer for exposure to hyperbaric pressure and 3.0 Tesla MRI.
* Participants who must travel to altitudes greater than 10,000 feet during chamber session intervention.
* Paratroopers who are unable to suspend activity during chamber exposures.
* An individual who has had refractive eye surgery within the last 90 days.
* Any brain injury not of traumatic etiology, such as stroke or drug-induced coma.
* Heart failure with ejection fraction < 50% (due to increased risk for precipitating acute lung edema during exposure to HBO2).
* Emphysema, chronic bronchitis, or bullous lung disease (due to risk for pulmonary barotrauma during hyperbaric decompression).
* Asthma not well controlled.

An individual with any of the following characteristics will be excluded from this study based on confounding of the outcome measures:

* Those who are unable to participate fully in outcome assessments unless randomization is reviewed and approved (in writing) by the study director.
* Vision uncorrectable to 20/50 (monocular vision acceptable).
* Dynavision within 30 days of screening.
* Deafness in both ears defined as 90 dB HL or greater, through the speech frequencies of each of 500 Hz, 1 kHz, 2 kHz and 4 kHz in each ear; this is determined by a baseline measurement of pure tone air conduction thresholds.
* Participant self-report or documented diagnosis of psychiatric disorders in the medical record within the last year of any of the following: schizophrenia, dissociative disorder, or bipolar disease.
* Anxiety or claustrophobia precluding participation in the hyperbaric chamber sessions or neuroimaging procedures.
* Verifiable neurodegenerative disease (e.g., Alzheimer's disease, multiple sclerosis, senile dementia).
* Presence of chronic debilitating disease (e.g., end-stage renal disease, end-stage liver disease, diabetes with sequelae).
* Documented unresolved anemia, with anemia defined as hematocrit less than 30%.
* History, by self-report, of receiving therapeutic ionizing radiation to the head.
* Foreign material in head that would interfere with brain imaging (e.g., MRI or computed tomography [CT]), unless randomization has been cleared by the study director.
* Foreign (unknown composition) or metallic/ferromagnetic material within the individual that poses risk from MRI, unless randomization has been cleared by the study director.
* History, by self report, of illicit drug use, except remote (prior to military enlistment) non-habitual (habitual is considered greater than weekend) use of marijuana.
* History, by self report or medical record in the last year, of alcohol abuse. Prospective participants who have been sober for the last 90 days prior to screening may be eligible based on the site principal investigator determination.
* Current positive urine test for an illicit substance(s).
* Any condition or use of prescribed medication in which, in the opinion of the investigator, participation in this study would impact the safety of the individual.
* Brain injury of moderate or severe degree: duration of loss of consciousness at the time of injury greater than 30 minutes, duration of post-traumatic amnesia greater than 24 hours, or brain injury of a penetrating etiology.
* Any lifetime history of penetrating brain injury.
* Active malignancy, prior malignancy (except basal cell carcinoma) within the last 5 years, or any prior treatment with bleomycin (trade name Blenoxane). Prior treatment with doxorubicin (trade name Adriamycin) is acceptable as long as an echocardiography following treatment is normal.
* Unable to abstain from caffeine or tobacco products for at least a 2-hour interval.
* Concurrent enrollment in an alternate interventional trial.
* Unable or unwilling to cease participation in sports in which another head injury is likely (e.g., mixed martial arts, boxing) during the study period.
* Diagnosis of Meniere's disease by self-report or medical record evidence within one year.
* Pre-TBI history of significant dizziness (lasting more than 1 day).

A prospective participant with any of the following characteristics will be excluded from this study to protect blinding:

* Prior treatment with HBO2 for TBI or PCS.
* Prior HBO2 treatment for indications other than TBI or PCS within the last 3 months.
* Experienced hyperbaric chamber inside attendant (anyone deemed to have experience with hyperbaric pressurization that could compromise their blind to allocation).
* Technical, military, or occupational divers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindell Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (5):
- United States (5):
  - Outcomes Assessment Center, Evans Army Community Hospital, Colorado Springs, Colorado
  - Evans Army Community Hospital / Hyperbaric Medicine Complex, Fort Carson, Colorado
  - Camp Lejeune, Jacksonville, North Carolina
  - Joint Base Lewis-McChord, Fort Lewis, Washington
  - TBI Program/HBO2 Research Program Madigan Healthcare system, Tacoma, Washington

REFERENCES:
- [Derived] Weaver LK, Churchill S, Wilson SH, Hebert D, Deru K, Lindblad AS. A composite outcome for mild traumatic brain injury in trials of hyperbaric oxygen. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):341-352. PMID 31394603
- [Derived] Churchill S, Deru K, Weaver LK, Wilson SH, Hebert D, Miller RS, Lindblad AS. Adverse events and blinding in two randomized trials of hyperbaric oxygen for persistent post-concussive symptoms. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):331-340. PMID 31394602
- [Derived] Hart BB, Wilson SH, Churchill S, Deru K, Weaver LK, Minnakanti M, Lindblad AS. Extended follow-up in a randomized trial of hyperbaric oxygen for persistent post-concussive symptoms. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):313-327. PMID 31394601
- [Derived] Wetzel PA, Lindblad AS, Mulatya C, Kannan MA, Villmar Z, Gitchel GT, Weaver LK. Eye tracker outcomes in a randomized trial of 40 sessions of hyperbaric oxygen or sham in participants with persistent post concussive symptoms. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):299-311. PMID 31394600
- [Derived] Walker JM, Mulatya C, Hebert D, Wilson SH, Lindblad AS, Weaver LK. Sleep assessment in a randomized trial of hyperbaric oxygen in U.S. service members with post concussive mild traumatic brain injury compared to normal controls. Sleep Med. 2018 Nov;51:66-79. doi: 10.1016/j.sleep.2018.06.006. Epub 2018 Jun 30. PMID 30099354
- [Derived] Wetzel PA, Lindblad AS, Raizada H, James N, Mulatya C, Kannan MA, Villamar Z, Gitchel GT, Weaver LK. Eye Tracking Results in Postconcussive Syndrome Versus Normative Participants. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):4011-4019. doi: 10.1167/iovs.18-23815. PMID 30098189
- [Derived] Meehan A, Searing E, Weaver LK, Lewandowski A. Baseline vestibular and auditory findings in a trial of post-concussive syndrome. Undersea Hyperb Med. 2016 Aug-Sept;43(5):567-584. PMID 28771392
- [Derived] Wilson SH, Weaver LK, Lindblad AS. Neuropsychological assessments in a hyperbaric trial of post-concussive symptoms. Undersea Hyperb Med. 2016 Aug-Sept;43(5):585-599. PMID 28768075
- [Derived] Walker JM, James NT, Campbell H, Wilson SH, Churchill S, Weaver LK. Sleep assessments for a mild traumatic brain injury trial in a military population. Undersea Hyperb Med. 2016 Aug-Sept;43(5):549-566. PMID 28768073
- [Derived] Mirow S, Wilson SH, Weaver LK, Churchill S, Deru K, Lindblad AS. Linear analysis of heart rate variability in post-concussive syndrome. Undersea Hyperb Med. 2016 Aug-Sept;43(5):531-547. PMID 28768072
- [Derived] Williams CS, Spitz MC, Foley JF, Weaver LK, Lindblad AS, Wierzbicki MR. Baseline EEG abnormalities in mild traumatic brain injury from the BIMA study. Undersea Hyperb Med. 2016 Aug-Sept;43(5):521-530. PMID 28768071
- [Derived] Williams CS, Weaver LK, Lindblad AS, Kumar S, Langford DR. Baseline neurological evaluations in a hyperbaric trial of post-concussive syndrome. Undersea Hyperb Med. 2016 Aug-Sept;43(5):511-519. PMID 28768070
- [Derived] Weaver LK, Chhoeu A, Lindblad AS, Churchill S, Wilson SH. Hyperbaric oxygen for mild traumatic brain injury: Design and baseline summary. Undersea Hyperb Med. 2016 Aug-Sept;43(5):491-509. PMID 28768069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from military sites from Sept 2012 to May 2014.
Period: Overall Study
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Started | 36 | 35
Completed | 36 | 32
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — drug use | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres) | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (8.3) | 30.8 (5.5) | 32.8 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 36 | 34 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 2 | 2 | 4
  White | 30 | 28 | 58
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 35 | 71
Education [Count of Participants; unit: Participants]
  Less than high school diploma | 0 | 0 | 0
  High school diploma | 7 | 6 | 13
  Some college | 13 | 23 | 36
  College degree | 11 | 5 | 16
  Graduare degree | 5 | 1 | 6
Military Status [Count of Participants; unit: Participants]
  Active duty | 35 | 33 | 68
  Veteran | 1 | 2 | 3
Time From Most Recent Qualifying Mild Traumatic Brain Injury (mTBI) [Mean (Standard Deviation); unit: months] | 25.6 (17.1) | 25.5 (15.4) | 25.6 (16.2)
Most Recent Qualifying mTBI 3 Months to 1 Year [Count of Participants; unit: Participants]
  3 months to 1 year | 12 | 8 | 20
  >1year to 5 years | 24 | 27 | 51
Number of Lifetime mTBIs [Mean (Standard Deviation); unit: mTBIs] | 3.6 (3.2) | 3.7 (2.3) | 3.6 (2.8)
Lifetime mTBI History [Count of Participants; unit: Participants]
  Blast injuries | 15 | 8 | 23
  Blunt force head injuries only | 7 | 7 | 14
  Combination of blast and blunt force injuries | 14 | 20 | 34
Most Recent Qualifying Injury [Count of Participants; unit: Participants]
  Blast injury | 23 | 23 | 46
  Blunt force head injury | 13 | 12 | 25
Military Rank [Count of Participants; unit: Participants]
  E1-E10 | 31 | 35 | 66
  O-1 to O-10/W-1 to W-5 | 5 | 0 | 5
Military Branch [Count of Participants; unit: Participants]
  Army | 27 | 28 | 55
  Marines | 7 | 5 | 12
  Navy, Air Force, and Coast Guard | 2 | 2 | 4
Number of Combat Deployments [Mean (Standard Deviation); unit: deployments] | 3.4 (2.8) | 2.2 (1.7) | 2.8 (2.4)
Common Medication Usage [Number; unit: participants]
  SSRI/SNRIs | 12 | 10 | 22
  Hypnotic or sleep aid | 16 | 15 | 31
  Daily pain medication | 22 | 21 | 43
  Episodic migraine medication | 16 | 14 | 30
  Fish oil or omega-3 fatty acid | 9 | 8 | 17
Common Alternative Therapy Usage [Number; unit: participants]
  Psychotherapy | 12 | 7 | 19
  Counseling | 16 | 12 | 28
  Physical therapy | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment-Emergent Adverse Events
Description: Safety was evaluated in-person during the first 3 months and at month 6, and via telephone follow-up calls at months 4, 5, and 7-12. Extended annual follow-up continued for up to 36 months through January 2016.
Time Frame: months 3, 6, 4, 5 and 7-12. Extended f/u up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
Participants
  Barotitis media | 13 | 5
  Sinus barotrauma | 5 | 3
  Contusion | 3 | 3
  Ligament sprain | 0 | 5
  Muscle strain | 1 | 3
  Upper respiratory tract infection | 13 | 9
  Gastroenteritis | 1 | 5
  Sinusitis | 3 | 4
  Nasopharyngitis | 3 | 2
  Arthralgia | 4 | 2
  Back pain | 3 | 2
  Neck pain | 0 | 4
  Dizziness | 5 | 1
  Headache | 4 | 2
  Nasal congestion | 5 | 3
  Dyspnea | 4 | 1
  Epistaxis | 2 | 2
  Sinus congestion | 2 | 2
  Eye disorders | 10 | 7
  Nausea | 4 | 1
  Suicidal ideation | 2 | 2
  Rash | 0 | 3
  Investigations | 4 | 3
  Vertigo | 3 | 3
  General and administration site conditions | 3 | 1
  Metabolism and nutrition disorders | 3 | 2
  Renal and urinary disorders | 3 | 0
  Vascular disorders | 3 | 0
  Congenital, familial and genetic disorders | 1 | 0
  Endocrine disorders | 1 | 0
  Hepatobiliary disorders | 1 | 0
  Immune system disorders | 0 | 1
  Neoplasms benign, malignant and unspecified | 0 | 1

2. Primary Outcome: Summary of Study Intervention-Related Adverse Events
Description: as for outcome 1
Time Frame: months 3, 6, 4, 5 and 7-12. Extended f/u up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
Participants
  Barotitis media | 11 | 5
  Sinus barotrauma | 5 | 4
  Dizziness | 1 | 1
  Headache | 1 | 2
  Somnolence | 1 | 1
  Dyspnea | 2 | 0
  Hyperventilation | 1 | 0
  Anxiety | 1 | 0
  Myopia | 1 | 1
  Eye pruritus | 0 | 1
  Vertigo | 1 | 1

3. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ, RPQ3 and RPQ13) - Baseline (ITT Population)
Description: RPQ/RPQ-3 was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-3 ranges from 0-12 and access a subset of symptoms. RPQ-13 ranges from 0-52 and access's 13 remaining symptoms. Analyses of the RPQ-3 and RPQ-13 domain scores are presented separately. For each of the RPQ-3, RPQ-13, and RPQ total scales, the scores were derived by totaling the corresponding question scores for each domain.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  RPQ Total Score | 34.8 (13.1) | 28.2 (13.5)
  RPQ-3 Score | 5.8 (2.9) | 4.5 (2.6)
  RPQ-13 Score | 29.0 (11.0) | 23.7 (11.4)

4. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ, RPQ3 and RPQ13) - Baseline (Per Protocol (PP) Population)
Description: as for outcome 3
Time Frame: Baseline
Population: PP was defined as subs who completed 20 chamber sessions and week13 f/u. PP was also restricted to subs who didn't report illicit drug use following randomization. 67 subs satisfied the PP, 35/36 HBO2 and 32/35 sham. 4 were excluded from the PP population, 3 excluded because they completed <20 sessions,1 because of illicit drug use during study.
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  RPQ Total Score | 34.7 (13.3) | 27.3 (12.9)
  RPQ-3 Score | 5.8 (2.9) | 4.5 (2.5)
  RPQ-13 Score | 28.9 (11.1) | 22.8 (11.0)

5. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ) - Change From Baseline (ITT Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. The scores were derived by totaling the corresponding question scores for each domain and it's change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: 1 subject in HBO2 missed the 6 month visit and 2 subjects missed the 12 month visit. 1 subject in the sham missed the week 13 visit and, 1 subject missed the month 6 visit and 3 subjects withdrew by month 12
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Week 13 change score | -0.7 (14.6) | 5.8 (12.4)
  Month 6 change score: number analyzed (Participants) | 35 | 32
  Month 6 change score | -4.3 (14.0) | 2.6 (11.6)
  Month 12 change score: number analyzed (Participants) | 34 | 31
  Month 12 change score | 5.7 (14.7) | 5.5 (12.4)

6. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ3) - Change From Baseline (ITT Population)
Description: RPQ-3 was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-3 ranges from 0-12 and access a subset of symptoms. Analyses of the RPQ-3 domain scores are presented separately. For the RPQ-3 total scales, the scores were derived by totaling the corresponding question scores for each domain and it's change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Week 13 change score | -0.3 (2.7) | 1.2 (2.2)
  Month 6 change score: number analyzed (Participants) | 35 | 32
  Month 6 change score | -1.4 (2.7) | 0.3 (2.2)
  Month 12 change score: number analyzed (Participants) | 35 | 31
  Month 12 change score | 0.5 (2.9) | 0.5 (2.6)

7. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ13) - Change From Baseline (ITT Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-13 ranges from 0-52 and access's 13 remaining symptoms. Analyses of the RPQ-13 domain scores are presented separately. For RPQ-13 total scales, the scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Week 13 change score | -0.4 (12.3) | 4.7 (11.1)
  Month 6 change score: number analyzed (Participants) | 35 | 32
  Month 6 change score | -3.0 (11.9) | 2.3 (9.9)
  Month 12 change score: number analyzed (Participants) | 34 | 31
  Month 12 change score | 5.2 (12.7) | 5.0 (10.4)

8. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ) - Change From Baseline (Per Protocol (PP) Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-3 ranges from 0-12 and access a subset of symptoms. For the RPQ total scales, the scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Week 13 change score | -1.0 (14.7) | 6.1 (12.6)
  Month 6 change score: number analyzed (Participants) | 35 | 31
  Month 6 change score | -4.3 (14.0) | 3.2 (11.3)
  Month 12 change score: number analyzed (Participants) | 33 | 30
  Month 12 change score | 5.8 (14.9) | 5.5 (12.6)

9. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ3) - Change From Baseline (Per Protocol (PP) Population)
Description: RPQ/RPQ-3 was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-3 ranges from 0-12 and access a subset of symptoms. For the RPQ-3total scale, the scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Week 13 change score | -0.4 (2.8) | 1.2 (2.3)
  Month 6 change score: number analyzed (Participants) | 35 | 31
  Month 6 change score | -1.4 (2.7) | 0.3 (2.2)
  Month 12 change score: number analyzed (Participants) | 34 | 30
  Month 12 change score | 0.4 (2.9) | 0.5 (2.7)

10. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ13) - Change From Baseline (Per Protocol (PP) Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". RPQ-13 ranges from 0-52 and access's 13 remaining symptoms. Analyses of the RPQ-13 domain scores are presented separately. The scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to week 13, Months 6 and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Week 13 change score | -0.7 (12.4) | 4.9 (11.2)
  Month 6 change score: number analyzed (Participants) | 35 | 31
  Month 6 change score | -3.0 (11.9) | 2.9 (9.5)
  Month 12 change score: number analyzed (Participants) | 33 | 30
  Month 12 change score | 5.4 (12.8) | 5.1 (10.6)

11. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ) - Change From Baseline: 24 and 36 Months (ITT Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. For the RPQ total scales, the scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to 24 months and 36 months
Population: HBO2: 25 subs consented to 24 and 36 month f/u; 23 subs completed month 24 and 9 completed month 36; 2 subs missed 24 month visit.
  Sham: 17 subs consented to 24 and 36 month f/u. 17 completed month 24 and 5 completed month 36
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Baseline to 24 months: number analyzed (Participants) | 20 | 15
  Baseline to 24 months | 1.2 (18.5) | 2.9 (11.9)
  Baseline to 36 months: number analyzed (Participants) | 8 | 5
  Baseline to 36 months | 1.4 (9.0) | 4.6 (19.6)

12. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ3) - Change From Baseline: 24 and 36 Months (ITT Population)
Description: RPQ-3 was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-3 ranges from 0-12 and access a subset of symptoms. Analyses of the RPQ-3 domain scores are presented separately. For the RPQ-3 total scales, the scores were derived by totaling the corresponding question scores for each domain and change from baseline.
Time Frame: Baseline to 24 months and 36 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Baseline to 24 months: number analyzed (Participants) | 21 | 16
  Baseline to 24 months | -0.2 (3.2) | -0.1 (2.7)
  Baseline to 36 months: number analyzed (Participants) | 9 | 5
  Baseline to 36 months | -0.9 (2.9) | 0.8 (3.0)

13. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ13) - Change From Baseline: 24 and 36 Months (ITT Population)
Description: as for outcome 7
Time Frame: Baseline to 24 months and 36 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 36 | 35
RPQ scores
  Baseline to 24 months: number analyzed (Participants) | 20 | 15
  Baseline to 24 months | 1.4 (16.1) | 3.0 (9.5)
  Baseline to 36 months: number analyzed (Participants) | 8 | 5
  Baseline to 36 months | 2.0 (7.5) | 3.8 (16.8)

14. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ) - Change From Baseline (Per Protocol (PP) Population)
Description: as for outcome 11
Time Frame: Baseline to month 24 and month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Baseline to month 24: number analyzed (Participants) | 20 | 15
  Baseline to month 24 | 1.2 (18.5) | 2.9 (11.9)
  Baseline to month 36: number analyzed (Participants) | 8 | 5
  Baseline to month 36 | 1.4 (9.0) | 4.6 (19.6)

15. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ3) - Change From Baseline (Per Protocol (PP) Population)
Description: as for outcome 12
Time Frame: Baseline to month 24 and month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Baseline to month 24: number analyzed (Participants) | 21 | 16
  Baseline to month 24 | -0.2 (3.2) | -0.1 (2.7)
  Baseline to month 36: number analyzed (Participants) | 9 | 5
  Baseline to month 36 | -0.9 (2.9) | 0.8 (3.0)

16. Secondary Outcome: Presence of Post Concussion Symptoms Following Traumatic Brain Injury Using The Rivermead Post-Concussion Symptom Questionnaire (RPQ13) - Change From Baseline (Per Protocol (PP) Population)
Description: RPQ was created to measure the severity of post-concussion symptoms following traumatic brain injury. Scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature. The RPQ scale includes 16 common post-concussion symptom items whose responses range from "0= Not experienced at" to "4= A severe problem". Total range is 0 to 64. RPQ-13 ranges from 0-52 and access's 13 remaining symptoms. Analyses of the RPQ-13 domain scores are presented separately. For RPQ-13 total scales, the scores were derived by totaling the corresponding question scores for each domain change from baseline.
Time Frame: Baseline to month 24 and month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: RPQ scores
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
Number analyzed (Participants) | 35 | 32
RPQ scores
  Baseline to month 24: number analyzed (Participants) | 20 | 15
  Baseline to month 24 | 1.4 (16.1) | 3.0 (9.5)
  Baseline to month 36: number analyzed (Participants) | 8 | 5
  Baseline to month 36 | 2.0 (7.5) | 3.8 (16.8)

ADVERSE EVENTS:
Time Frame: Safety was evaluated in-person during the first 3 months and at month 6, and via telephone follow-up calls at months 4, 5, and 7-12. Extended annual follow-up continued for up to 36 months through January 2016.
Arm/Group | HBO2 at 1.5 Atomspheres Absolute (ATA) | Sham Control (1.2 Atomspheres)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 5/36 | 3/35
Other Adverse Events (participants affected / at risk) | 35/36 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBO2 at 1.5 Atomspheres Absolute (ATA) (N=36) | Sham Control (1.2 Atomspheres) (N=35)
Post-traumatic stress disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBO2 at 1.5 Atomspheres Absolute (ATA) (N=36) | Sham Control (1.2 Atomspheres) (N=35)
Barotitis media (Injury, poisoning and procedural complications) | 13 (20) | 6 (8)
Sinus barotrauma (Injury, poisoning and procedural complications) | 5 (10) | 4 (9)
Contusion (Injury, poisoning and procedural complications) | 6 (8) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Mucsle strain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 16 (18) | 10 (13)
Gastroenteritis (Infections and infestations) | 1 (1) | 6 (7)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 6 (7) | 1 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2)
Eye disorders (Eye disorders) | 11 (14) | 7 (10)
Vertigo (Ear and labyrinth disorders) | 3 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3)
Investigations (Investigations) | 5 (7) | 3 (4)
General disorders and administration site conditions (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Vascular disorders (Vascular disorders) | 5 (6) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 3 (4) | 0 (0)
Immune system disorders (Immune system disorders) | 1 (1) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No